CLINICAL TRIAL: NCT01476644
Title: A Prospective, Longitudinal, Observational Cohort Study Examining How Glaucoma Affects Quality of Life and Visual Function Over a 4-Year Period
Brief Title: How Has Glaucoma Affected Your Quality of Life?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, George L. Spaeth MD, Principal Investigator, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB#11-128
Record Dates: First submitted 2011-10-31; First posted 2011-11-22 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Glaucoma; Quality of Life
Keywords: Health related quality of life; Clinical measures of vision
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: A prospective, longitudinal,observational cohort study to investigate how glaucoma affects patients' quality of life and visually-related function. Annual visits included (1) Clinical evaluation: a slit lamp examination, fundoscopy, intraocular pressure measurement, visual field examination, spectral domain optical coherence tomography, Pelli-Robson Contrast Sensitivity test and the Spaeth-Richman Contrast Sensitivity test; (2) a performance based measure: the Compressed Assessment of Ability Related to Vision; and (3) Subjective measures of vision-related quality of life (the National Eye Institute Visual Functioning Questionnaire 25 and the Modified Glaucoma Symptom Scale).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glaucoma Patients (Other): Moderate glaucoma patients with a minimum 2-year diagnosis of primary open-angle glaucoma, chronic primary angle-closure glaucoma or pseudoexfoliation glaucoma were included to complete annual visits over a 4 year period. Each visit included (1) Clinical evaluation: a slit lamp examination, fundoscopy, intraocular pressure measurement, visual field examination, spectral domain optical coherence tomography, Pelli-Robson Contrast Sensitivity test and the Spaeth-Richman Contrast Sensitivity test; (2) a performance based measures: the Compressed Assessment of Ability Related to Vision; and (3) Subjective measures of vision-related quality of life (VRQoL) (the National Eye Institute Visual Functioning Questionnaire 25 and the Modified Glaucoma Symptom Scale).
  Interventions: Other: Clinical evaluation; Other: Performance based measures; Other: Subjective measures of vision-related quality of life

INTERVENTIONS:
Other: Clinical evaluation — Biomicroscopy (look at front of eye), ophthalmoscopy (look at back of eye), visual acuity, visual fields, intraocular pressure, spectral domain optical coherence tomography, Pelli-Robson and the Spaeth-Richman Contrast Sensitivity tests
  Other Names: Ophthalmic examination
Other: Performance based measures — Compressed Assessment of Ability Related to Vision (CAARV) items include: 1) computerized motion detection; 2) recognizing facial expressions; 3) reading street signs; and 4) finding objects in a room
  Other Names: Compressed Assessment of Ability Related to Vision
Other: Subjective measures of vision-related quality of life — National Eye Institute Visual Functioning Questionnaire 25 (NEI-VFQ-25) includes a series of questions pertaining to vision or feelings about a vision condition and the Modified Glaucoma Symptom Scale (MGSS) includes a series of questions pertaining to eye comfort.
  Other Names: Visual Functioning Questionnaire; Modified Glaucoma Symptom Scale

SUMMARY:
Hypothesis 1: Self-reported health-related quality of life decreases as vision impairment worsens in subjects with glaucoma.

Hypothesis 2: Changes in health-related quality of life are associated with changes in clinical measures of vision and performance-based measures of visual function.

DETAILED DESCRIPTION:
You are being asked to participate in this research study because you have glaucoma, which is the second leading cause of blindness in the world and accounts for 15% of blindness worldwide. Vision loss caused by glaucoma can significantly worsen your health-related quality of life. Despite the fact that glaucoma has such a big impact on a large number of people, research examining the long-term effects of glaucoma-related vision loss on one's quality of life is scarce.

The purpose of this study is to look at the long-term effect of this condition on your quality of life so that we may gain valuable information about what factors influence the quality of life of people with glaucoma. To participate in this study, you will need to allow us to perform clinical tests on your eyes, to self-report your well-being and health-related quality of life, and to let us know how well you perform your daily life activities.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 2-year diagnosis of primary open-angle glaucoma, chronic primary angle-closure glaucoma or exfoliation glaucoma
* Disk Damage Likelihood Scale stages 5 through 8 with visual field loss
* Age between 21 and 80 years
* Able to understand and speak English

Exclusion Criteria:

* Unlikely to be available for annual ocular examination and reassessment across a 4-year period
* Neurological or musculoskeletal problems that would influence performance on activities of daily living
* Cognitively impaired, as assessed by a face-to-face Mini-Mental State Examination
* Incisional eye surgery within the past three months
* Laser therapy within the previous month
* Any cause for visual reduction other than glaucoma
* Any medical condition which in the investigator's opinion would preclude the subject from providing reliable and valid data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Glaucoma Service, Wills Eye Institute
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Erdem E, Wizov S, Kayak N, Wei H, Spaeth GL. Quality of life measures in moderate glaucoma: study design and methodology. Abstract submitted, Association for Research in Vision and Ophthalmology, Dec 2012.
- [Background] Ekici F, Sun Y, Taranum S, Martinez P, Erdem E, Nayak N, Wizov SS, Waisbourd M, Spaeth GL. Relationship between baseline clinical characteristics and vision-related quality of life in patients with glaucoma. ARVO Poster 176-A0363 May 2014.
- [Background] Gogte P., Hark LA., Spaeth E., Richman J., Wizov SS., Waisbourd M., Spaeth GL. Contrast Sensitivity - A Meaningful Way to Assess Health Related Quality of Life and Ability to Perform Daily Activities in Glaucoma Patients. ARVO Poster 2097-A0004 May 2015.
- [Background] Waisbourd M., Gogte P., Richman J., Spaeth E., Dai Y., Wizov SS., Hark LA., Spaeth GL. Comparative Results with Regards to Humphrey Visual Fields and the SPARCS Contrast Sensitivity Test in Patients with Glaucoma. AOS meeting April 2015.
- [Result] Waisbourd M, Parker S, Ekici F, Martinez P, Murphy R, Scully K, Wizov SS, Hark LA, Spaeth GL. A prospective, longitudinal, observational cohort study examining how glaucoma affects quality of life and visually-related function over 4 years: design and methodology. BMC Ophthalmol. 2015 Aug 1;15:91. doi: 10.1186/s12886-015-0088-x. PMID 26231376
- [Result] Ekici F, Loh R, Waisbourd M, Sun Y, Martinez P, Nayak N, Wizov SS, Hegarty S, Hark LA, Spaeth GL. Relationships Between Measures of the Ability to Perform Vision-Related Activities, Vision-Related Quality of Life, and Clinical Findings in Patients With Glaucoma. JAMA Ophthalmol. 2015 Dec;133(12):1377-85. doi: 10.1001/jamaophthalmol.2015.3426. PMID 26425961
- [Result] Sun Y, Lin C, Waisbourd M, Ekici F, Erdem E, Wizov SS, Hark LA, Spaeth GL. The Impact of Visual Field Clusters on Performance-based Measures and Vision-Related Quality of Life in Patients With Glaucoma. Am J Ophthalmol. 2016 Mar;163:45-52. doi: 10.1016/j.ajo.2015.12.006. Epub 2015 Dec 14. PMID 26701273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Moderate glaucoma subjects recruited from the Glaucoma Service at Wills Eye Hospital, Philadelphia, Pennsylvania between May 2012 and May 2014 for an observational longitudinal study. One baseline and four annual visits were performed.
Groups:
- Participants With Moderate Glaucoma: Participants with moderate glaucoma as defined by a disc damage likelihood scale (DDLS range 1 to 9) of the optic nerve between 5 and 8 in at least one eye. One on the DDLS corresponds to healthy optic nerve; 9 is advanced glaucoma damage.
Period: Overall Study
Arm/Group | Participants With Moderate Glaucoma
Started | 161
Completed | 122
Not Completed | 39
Not completed — Death | 5
Not completed — moved to another state | 2
Not completed — Lost to Follow-up | 19
Not completed — Withdrawal by Subject | 13

BASELINE CHARACTERISTICS:
Groups:
- Cohort: Moderate glaucoma with a DDLS (optic disc damage likelihood scale range 1-10 with 10 being worse ) between 5 and 8 in at least one eye.
Arm/Group | Cohort
Number analyzed (Participants) | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 159
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 52
  White | 96
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161
NEI-VFQ 25 [Mean (Standard Deviation); unit: units on a scale] — National Eye Institute - Visual Function Questionnaire 25 regarding quality of life related to vision measures participants perception of how well they are managing with their level of vision. Questionnaire scores range from 0 to 100 with 0 representing significant difficulties and 100 equals no difficulties at all.
  units on a scale | 83.5 (14.3)
MGSS [Mean (Standard Deviation); unit: units on a scale] | 83.7 (13.1)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life With NEI VFQ-25
Description: National Eye Institute Visual Function-25 questionnaire (NEI VFQ-25) is a measurement of patients perception of their visually related quality of life. Patients select answers from multiple choice lists of responses. Values are re-coded and converted to a scale of 0 to 100 where 0 is extreme difficulty and 100 is no difficulty at all (or best quality of life). Data from visits 2 through 5.
Time Frame: 2 hours at each annual visit, visits 2 through 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cohort: Moderate glaucoma participants based on a DDLS (disc damage likelihood scale, a grade of the health of the optic nerve) between 5 and 8 in at least one eye. DDLS score ranges from 1 to 10 with 10 being worst optic nerve.
Arm/Group | Cohort
Number analyzed (Participants) | 161
units on a scale
  Visit 2 | 82.9 (13.6)
  Visit 3 | 82.7 (14.7)
  Visit 4 | 82.8 (13.5)
  Visit 5 | 83.0 (14.8)

2. Secondary Outcome: Eye Comfort With MGSS
Description: Modified Glaucoma Symptom Scale (MGSS), is patient perception of their eyes comfort. Ten ocular complaints often associated with glaucoma each have a four level score (1 signifying very bothersome; 4 represents absence of problems). Scores from 10 questions are added and range from 0 to 100 where 0 represents significant discomfort and 100 represents no problems at all. The final MGSS score is an unweighted average of responses to 10 items, averaged between the 2 eyes. Data from visits 2 through 5.
Time Frame: 2 hours at each annual visit, visits 2 through 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cohort: All participants with moderate glaucoma measured by a DDLS (disc damage likelihood scale) between 5 and 8 in at least one eye agreed to the study.
Arm/Group | Cohort
Number analyzed (Participants) | 161
units on a scale
  Visit 2 | 84.0 (12.6)
  Visit 3 | 84.5 (13.0)
  Visit 4 | 86.1 (10.9)
  Visit 5 | 85.0 (13.9)
Statistical Analysis 1: Comparison: Cohort; Test type: Superiority or Other; p < 0.01, Regression, Linear

ADVERSE EVENTS:
Time Frame: 1 visit per year over 4 years
Groups:
- Cohort: Moderate glaucoma as confirmed by a DDLS (disc damage likelihood scale, optic nerve health) between 5 and 8 in at least one eye. DDLS range 1 to 10 with 10 being worse optic nerve damage.
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 5/161
Serious Adverse Events (participants affected / at risk) | 5/161
Other Adverse Events (participants affected / at risk) | 0/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort (N=161)
Death (Investigations) | 5 (5) — Events leading to deaths during participation in this four year observational trial were not study related. All deaths were reported to Wills Eye Hospital Institutional Review Board (IRB) before January 2017. No study intervention; no relationship.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No